CLINICAL TRIAL: NCT05821218
Title: Evaluation of the Sacroiliac Joints of People With Chronic Low Back Pain From a Chiropractic Perspective
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Erdal Beken, Principal Investigator, Bahçeşehir University
Other Study IDs: Chiropractic Perspective
Record Dates: First submitted 2023-03-24; First posted 2023-04-20 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Back Pain
Keywords: sacroiliac
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- back pain group: back pain group

SUMMARY:
Low back pain is a musculoskeletal problem that we commonly encounter in the clinic,which negatively affects the quality of life, reduces productivity and limits the ability to perform activities of daily living.

DETAILED DESCRIPTION:
The most common causes of low back pain are disc lesions and soft tissue injuries due to trauma, rheumatological disorders such as spondylosis, spinal stenosis and spondylolisthesis, ankylosing spondylitis and rheumatoid arthritis due to degenerative changes; osteoporosis, root disorders, and sacroiliac joint dysfunction

ELIGIBILITY:
Inclusion criteria;

* Volunteer
* Not undergoing surgery related to the lumbar region
* Cases without lumbar steroid injection in the last 3 months
* Not having visual and hearing loss
* Having low back pain
* Cases without neurological problems
* Cases without tumor and infection in the lumbar region
* Cases in which communication and cooperation are provided Exclusion criteria;
* Not having a musculoskeletal or neuromuscular disease that limits mobility,
* No upper extremity sequelae,
* Not volunteering

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bahçeşehir University
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-07-23 (Estimated)

PRIMARY OUTCOMES:
Leg Check Test | 1 day
  When a subject is lying prone or supine, emptying the pelvis, the feet are examined for the presence of a "short leg" or alignment asymmetry, often at the margin (heel-sole interface). Evidence has suggested that for most people, anatomical leg length disparity is not clinically relevant until the size reaches ~20 mm (~3/4"). It is a clinical test commonly used by chiropractors
Pressure Pain Threshold Measurement with Algometer | 1 day
  Pressure algometry is a semi-quantitative method used to localize sensitive areas, trigger points, abnormal sensitivity on muscles and bones, and evaluate pressure pain sensitivity in tissues. The dial is calibrated to 2.5 kg in 25 g divisions. The pressure applied by continuously pressing the disc 35 against the skin is to advance the pointer on the dial clockwise through the metal piston.
Oswestry Disability Index | one day
  Low back pain is one of the most common disorders that cause activity limitationIt has 16 questions and two subscales: physical activity and work. The physical activity section consists of 5 questions and the labor section consists of 11 questions. The questionnaire was a 7-point Likert type scale. In the answers given to the questionnaire, 0 points are given to the statement of "I don't agree at all" and 6 points to the statement of "I totally agree".
Patrick FABER Test: | 1 day
  The ipsilateral hip and knee joint of the participant in the supine position was flexed, and the heel was placed on the opposite knee. The test stresses the anterior sacroiliac ligaments and hip joint. It was accepted that the pain was felt in the sacroiliac joint region
Gaenslen Test | 1 day
  The participant was in the supine position on the examination table, with the lower extremity close to the evaluator hanging down from the bed, while the hip joint was brought to maximal hyperextension, while the hip and knee joints were passively brought to maximum flexion in the other lower extremity. The
Compression Test | 1 day
  The participant was positioned on their side, hips flexed to 45° and knees flexed to 90°. The evaluator applied a compression force from the superior iliac crest to the lower iliac crest behind the patient. This test stretches the posterior sacroiliac ligaments and compresses the anterior portion of the sacroiliac joint. The test was considered positive if there was pain in the sacroiliac joint.
The straight leg raise test | 1 day
  The straight leg raise test is known as the sciatic nerve stretch test. It has been reported that mobilization and stretching of the sciatic nerve occur from 30 degrees on.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No